CLINICAL TRIAL: NCT04997499
Title: Validation of a Video Teaching Tool for Adolescent Self Administration of Subcutaneous Depot-medroxyprogesterone
Brief Title: Adolescent Subcutaneous (SQ) Injection Video Validation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 00001518
Record Dates: First submitted 2021-07-20; First posted 2021-08-09 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Medication Compliance; Contraception; Self-Evaluation
Keywords: adolescent medication self-administration; subcutaneous depot-medroxyprogesterone; video instruction
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: Subjects will be current users of depot-medroxyprogesterone via intramuscular injection and will be asked to watch a video to instruct them on how to self administer a subcutaneous injection of the same medication
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Teaching video (Experimental): This is a single arm interventional study wherein the subjects enrolled will all participate in the study in the same way by watching the teaching video and then will be asked to self inject subcutaneous depot-medroxyprogesterone as per the protocol. All participants will then be asked to answer survey questions. All health care providers that participate in the study will likewise be asked to answer survey questions.
  Interventions: Behavioral: watch an instructional video

INTERVENTIONS:
Behavioral: watch an instructional video — watch instructional video and then perform self injection of subcutaneous depot-medroxyprogesterone based on the video teaching

SUMMARY:
This is a study to determine if a video that utilizes a peer to teach self administration of subcutaneous depot medroxyprogesterone is both effective and well accepted by adolescent patients who are already receiving ongoing treatment with depot medroxyprogesterone by a medical provider via an inter muscular injection. Self administration can be done at home and therefore offers an alternative to traveling to a medical office.

DETAILED DESCRIPTION:
Means of providing health education are rapidly evolving. Telemedicine has become an important modality to provide healthcare and improve access, and will likely be increasingly utilized beyond the COVID-19 pandemic. Telemedicine can effectively provide care and counseling to all age groups, including adolescents. Studies have demonstrated that over 80 percent of adolescents between the ages of 11 and 18 spend one to four hours a day online; searches for health-related information are common. Nevertheless, adolescents may face obstacles when previously familiar aspects of their medical care are abruptly moved online, particularly when discussing contraception. Although traditionally administered in the clinical space, injectable contraception has been shown to be attractive, effective, and well-tolerated by adolescents when subcutaneously self-administered, and can lead to improved continuation rates. The investigators have found that remotely teaching a patient how to self-administer a subcutaneous injection is challenging. The provider may be in a home office, and may not have access to the actual medication or the supplies to demonstrate technique. The patient may struggle to understand verbal instruction without a visual demonstration, resulting in ineffective medication administration. Instructional videos currently available online are not specific to adolescents who use self-administered injectable contraception. Peer education can be relatable and effective for adolescent patients. The investigators propose that self-administration of subcutaneous injectable contraception may be taught using a peer-to-peer video as a synchronous or asynchronous adjunct to consultation with the healthcare professional. Adolescents may be instructed to watch the video demonstration to help inform them about proper technique and ensure safe administration of their medication while at home. This study aims to validate an existing video as an effective teaching tool by assessing metrics such as clarity of the instructions, rate of error, and satisfaction with the video teaching method to the investigators' target population. The video was filmed in accordance with Tufts Medical Center Department of Marketing and Communications policies and the adolescent participant in the video was appropriately consented by a parent/guardian. The video was presented as an oral abstract at the North American Society for Pediatric and Adolescent Gynecology Annual Meeting in March 2021.

Procedure:

1. Clinic schedules for the medical providers on the research team will be reviewed in advance and any patient that is under the age of 20 and receiving depot-medroxyprogesterone will be contacted by telephone in advance to offer participation in the project.
2. The telephone call will follow the attached script. Two attempts will be made to call patients.
3. If subject is interested in participating, a prescription for the subcutaneous version of depot-medroxyprogesterone will be sent to their pharmacy to be picked up by the subject prior to the office visit.
4. Subjects under 18 will be instructed that they must be accompanied by a parent or guardian. At the office visit, written consent/assent will be obtained. 5. Subject will be shown the instructional video, which is approximately 3 minutes long. Subject may view as many times as subject chooses.

6. Once ready, the healthcare provider from the research team will observe, without giving verbal instruction, the subject self administer a subcutaneous depot-medroxyprogesterone injection.

7. If at any point the provider feels that the subject is not performing the injection safely or correctly the healthcare provider will intervene to ensure that the medication is given correctly, and this will be recorded within the REDCap survey.

8. After the injection is given, the subject will fill out the REDCap survey, and the study team member administering injection will input observational data into REDCap.

9. Subject will be asked to repeat another questionnaire in REDCap at the time of the next injection which will be scheduled for 12 weeks later. The next visit is as per standard of care scheduling (this medication is routinely administered at approximately 12-week intervals). If the subject comes into the same office for the injection, the survey will be filled out in person. If the subject does not come into the same office, a link to the follow-up REDCap survey will be emailed to the subject with instructions on how to access the survey. Email addresses will be confirmed at the time of the first visit, as is routine for medical care.

ELIGIBILITY:
Inclusion Criteria:

* assigned females at birth aged 19 years and younger
* must have previously received at least one injection of depot medroxyprogesterone

Exclusion Criteria:

* never received a prior dose of depot medroxyprogesterone.
* any history of self-administered injectable medication (either intramuscular or subcutaneous)
* inability to understand written or spoken English
* no parent or guardian to sign consent if under age 18
* inability to watch the instructional video
* cognitive impairment
* pregnancy
* ward of the state
* prisoner

Max Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Supervised self-injection | 12-18 months
  This measure is coded 1 if the patient successfully completes self-injection at the first session after watching the video. Otherwise, the measure is coded 0. Incomplete attempts, such preparing for but not completing the injection, will be coded 0.

SECONDARY OUTCOMES:
Sustained self-injection | 12-18 months
  This measure will be a count of self reported self injections in the 10-14 weeks following initial visit. This information will be collected through a self reported electronic REDCap survey that is administered once after the initial survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang CJ, Ma J, Zuckerman B, Car J. The Opportunities for Telehealth in Pediatric Practice and Public Health. Pediatr Clin North Am. 2020 Aug;67(4):603-611. doi: 10.1016/j.pcl.2020.03.001. PMID 32650856
- [Background] Strasburger VC, Jordan AB, Donnerstein E. Health effects of media on children and adolescents. Pediatrics. 2010 Apr;125(4):756-67. doi: 10.1542/peds.2009-2563. Epub 2010 Mar 1. PMID 20194281
- [Background] Park E, Kwon M. Health-Related Internet Use by Children and Adolescents: Systematic Review. J Med Internet Res. 2018 Apr 3;20(4):e120. doi: 10.2196/jmir.7731. PMID 29615385
- [Background] Kennedy CE, Yeh PT, Gaffield ML, Brady M, Narasimhan M. Self-administration of injectable contraception: a systematic review and meta-analysis. BMJ Glob Health. 2019 Apr 2;4(2):e001350. doi: 10.1136/bmjgh-2018-001350. eCollection 2019. PMID 31179026
- [Background] Williams RL, Hensel DJ, Fortenberry JD. Self-administration of subcutaneous depot medroxyprogesterone acetate by adolescent women. Contraception. 2013 Sep;88(3):401-7. doi: 10.1016/j.contraception.2012.11.019. Epub 2013 Jan 4. PMID 23294549
- [Background] Cameron ST, Glasier A, Johnstone A. Pilot study of home self-administration of subcutaneous depo-medroxyprogesterone acetate for contraception. Contraception. 2012 May;85(5):458-64. doi: 10.1016/j.contraception.2011.10.002. Epub 2011 Nov 12. PMID 22079602
- [Background] Patton GC, Sawyer SM, Santelli JS, Ross DA, Afifi R, Allen NB, Arora M, Azzopardi P, Baldwin W, Bonell C, Kakuma R, Kennedy E, Mahon J, McGovern T, Mokdad AH, Patel V, Petroni S, Reavley N, Taiwo K, Waldfogel J, Wickremarathne D, Barroso C, Bhutta Z, Fatusi AO, Mattoo A, Diers J, Fang J, Ferguson J, Ssewamala F, Viner RM. Our future: a Lancet commission on adolescent health and wellbeing. Lancet. 2016 Jun 11;387(10036):2423-78. doi: 10.1016/S0140-6736(16)00579-1. Epub 2016 May 9. No abstract available. PMID 27174304

DOCUMENTS (2):
  • Study Protocol (2021-07-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT04997499/Prot_000.pdf
  • Informed Consent Form (2021-07-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT04997499/ICF_001.pdf